CLINICAL TRIAL: NCT05348356
Title: A Phase 2 Trial of Nirogacestat in Patients With Recurrent Ovarian Granulosa Cell Tumors
Brief Title: Nirogacestat in Ovarian Granulosa Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIR-OGT-201
Record Dates: First submitted 2022-04-13; First posted 2022-04-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Granulosa-Stromal Tumor; Ovarian Granulosa Cell Tumor; Ovarian Cancer
MeSH Terms: conditions — Granulosa cell tumor of the ovary; Ovarian Neoplasms | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nirogacestat Open-Label (Experimental): Nirogacestat 150 mg by mouth, twice daily
  Nirogacestat oral tablet: Nirogacestat tablet
  Interventions: Drug: Nirogacestat

INTERVENTIONS:
Drug: Nirogacestat — nirogacestat oral tablet
  Other Names: PF-03084014

SUMMARY:
This phase 2 clinical trial will study the effectiveness of nirogacestat in ovarian granulosa cell tumors (OvGCTs). Nirogacestat is a gamma secretase inhibitor (GSI) which is hypothesized to decrease the growth and activity of ovarian granulosa tumors.

DETAILED DESCRIPTION:
Ovarian granulosa cell tumors (OvGCTs) represent 5-7% of all ovarian cancers (~1.5 to 2k newly diagnosed patients/year in the United States) and are the most common subtype of ovarian sex cord tumors (70%). Treatment of granulosa cell tumors with nirogacestat is expected to inhibit Notch-induced granulosa cell proliferation.

This is a multi-center, single-arm, Phase 2 open label treatment study to determine the efficacy, safety, tolerability, and pharmacokinetics of nirogacestat in adult participants with relapsed/refractory OvGCT. The participants will continue treatment until disease progression as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (unless the participants meet criteria for continued treatment) or unacceptable toxicity.

ELIGIBILITY:
Key Inclusion Criteria:

* Has histologically confirmed recurrent adult-type granulosa cell tumor of the ovary prior to first dose of study treatment
* Have documented radiological evidence of relapse after at least one systemic therapy that is not amenable to surgery, or radiation and have measurable disease by RECIST v1.1 criteria
* Have adequate bone marrow, renal and hepatic function as defined by screening visit laboratory values

Key Exclusion Criteria:

* Has signs of bowel obstruction requiring parenteral nutrition, malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of nirogacestat
* Has had a major cardiac or thrombo-embolic event within 6 months of signing informed consent
* Has abnormal QT interval at Screening, or has congenital or acquired long QT syndrome or a history of additional risk factors for Torsades de Pointes
* Has current or chronic history of liver disease or known hepatic or biliary abnormalities
* Has received bevacizumab treatment or other monoclonal antibody therapy with targeted anti-angiogenic activity for OvGCT within 28 days (or 5 half-lives, whichever is shorter) prior to the first dose of study treatment;
* Has received treatment for OvGCT including but not limited to the following within 28 days (or 5 half-lives, whichever is longer) prior to the first dose of study treatment: hormonal therapy, chemotherapy, immunotherapy, targeted therapy or any investigational treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2.5 years
  The proportion of participants with complete response (CR) + partial response (PR) assessed using RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Progression Free Survival at 6 months (PFS-6) | First day of cycle 7 (approximately 6 months after the first dose of study treatment). Each cycle is 28 days.
  The number of participants without progression according to RECIST v1.1 or death at 6 months.
Overall Survival | 2 years after first dose of study treatment
  The number of participants who have not died of any cause.
Participant reported ovarian cancer symptoms | At each study visit until study completion (estimated to be an average of 2.5 years)
  Change from baseline as measured by Functional Assessment of Cancer Therapy - Ovarian Symptom Index (FOSI).
Duration of Response | First day of every other cycle (each cycle is 28 days) for the first year, and then every 3 cycles thereafter until study completion (estimated to be an average of 2.5 years).
  The time from response (CR + PR using RECIST v.1.) to disease progression and/or death

CONTACTS AND LOCATIONS:
Locations (21):
- United States (16):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA-JCCC Dept. of OBGYN - Women's Health Clinical Research Unit, Los Angeles, California
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Women's Cancer Care, Covington, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - David C. Pratt Cancer Center, St Louis, Missouri
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Institute, New York, New York
  - Women's Cancer Center at Kettering, Kettering, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - UW/Fred Hutch Cancer Center, Seattle, Washington
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- Cross Cancer Institute, Edmonton, Alberta, Canada
- Poland (4):
  - Maria Sklodowska-Curie Bialystok Oncology Center, Bialystok
  - Jagiellonian Innovation Centre Clinical Research Centre, Krakow
  - University Teaching Hospital Poznan, Department of Oncological Gynaecology, Poznan
  - Maria Sklodowska-Curie National Institute of Oncology-National Research Institute, Clinic of Oncological Gynecology, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent patient-level data from completed clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.

DOCUMENTS (2):
  • Study Protocol (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT05348356/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT05348356/SAP_001.pdf